CLINICAL TRIAL: NCT02270372
Title: A Phase 1b Study of ONT 10 and Varlilumab in Patients With Advanced Ovarian Cancer or Breast Cancer
Brief Title: Study of ONT-10 and Varlilumab to Treat Advanced Ovarian or Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONT-10-104
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-08

CONDITIONS: Advanced Breast Carcinoma; Advanced Ovarian Carcinoma
Keywords: Advanced breast carcinoma; Advanced ovarian carcinoma; MUC1; vaccine; Phase 1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Combination (Experimental): The drug combination of ONT-10 and varilumab
  Interventions: Biological: ONT-10, Varlilumab combination

INTERVENTIONS:
Biological: ONT-10, Varlilumab combination — ONT-10 a liposomal synthetic glycopolypeptide MUC1 targeted antigen formulated with PET Lipid A adjuvant.
  Varlilumab is a recombinant, fully human mAb of the IgG1κ isotype that specifically binds human CD27.

SUMMARY:
This is a two-part Phase 1b, open-label study of ONT 10 administered in combination with varlilumab. Two different doses of varlilumab will be studied in combination with the single agent recommended dose of ONT 10. Intermediate and/or lower doses of varlilumab or ONT-10 may also be studied at the recommendation of the safety monitoring committee (SMC).

DETAILED DESCRIPTION:
This is a two-part Phase 1b, open-label study of ONT 10 administered in combination with varlilumab. Two different doses of varlilumab will be studied in combination with the single agent recommended dose of ONT 10. Intermediate and/or lower doses of varlilumab or ONT-10 may also be studied at the recommendation of the safety monitoring committee (SMC). Treatment will be administered in cycles of 12 weeks each. All patients will receive a single dose of cyclophosphamide on Day -3. During Cycle 1, patients will receive ONT-10 administered SC once per week for 8 weeks followed by ONT-10 once every 6 weeks starting with Cycle 2, in combination with varlilumab administered IV once every 3 weeks x 3 doses, and then once every 6 weeks for cycles 2 through 5.

Each cohort will enroll an initial group of 6 evaluable patients with either breast or ovarian carcinoma. Initial enrollment into a cohort will be staggered, with the first patient treated in any new cohort to be followed for a minimum of two weeks for the occurrence of Unacceptable Toxicity prior to enrollment of the remaining 5 patients. Subsequent enrollment into a cohort may then continue without a staggered schedule until 6 patients treated are considered evaluable. Up to 24 additional evaluable patients may be enrolled and treated in Part 2 at the RD of varlilumab and ONT-10 identified in Part 1, including approximately equal numbers of patients with breast carcinoma (n~12) and ovarian carcinoma (n~12). Treatment in Part 2 will follow the same schedule as in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age at the time of consent
2. Life expectancy of at least 6 months, in the opinion of the investigator
3. Have histologically confirmed breast or ovarian carcinoma
4. Have evidence of persistent, recurrent, or progressive disease for which there is no known or established treatment available with curative intent, after at least one course of systemic therapy for locally advanced or metastatic disease , including chemotherapy, targeted therapy (small molecule or antibody based), or hormonal therapy
5. Measurable or evaluable disease by RECIST 1.1
6. ECOG performed status of 0 or 1
7. Adequate hematologic function defined by:
8. WBC count ≥ 3.0 x 103 cells/µL
9. Lymphocyte count ≥ 0.8 x 103 cells/µL
10. Platelet count ≥ 75 x 103 /µL, and
11. Hemoglobin ≥ 9 g/dL
12. Have renal and hepatic function as defined by:
13. AST and ALT ≤ 2.5 X ULN
14. Total bilirubin ≤ 1.5 X ULN. Patients with elevated bilirubin known to be due to Gilbert's disease may be enrolled after approval from the medical monitor, and
15. Creatinine clearance ≥ 50 mL/min
16. If female of child bearing potential, have a negative pregnancy test at screening
17. If fertile male or female of child-bearing potential, agree to consistently use a highly effective method of birth control (including birth control pills, barrier device, or intrauterine device, abstinence or other methods prescribed by a licensed healthcare provider) from the time of consent through 70 days following the last dose of study drug
18. Patient or a legally authorized representative of a patient must be able and willing to sign informed consent document that has been approved by an IRB

Exclusion Criteria:

1. Has medical, social, or psychological factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures
2. Is pregnant, breastfeeding, or planning a pregnancy
3. Has received treatment with any systemic anticancer therapy, wide-field radiation, or experimental agent within 4 weeks of receiving cyclophosphamide on Day -3, with the exception of anticancer hormonal therapy, which may not be given within 2 weeks of receiving cyclophosphamide on Day -3. All residual toxicity related to prior anticancer therapies (excluding vitiligo, endocrinopathies on stable replacement therapy, alopecia and Grade 2 fatigue) must resolve to Grade 1 severity or less or return to baseline prior to receipt of study treatment.
4. Has received treatment with focal radiotherapy within 2 weeks, or radiopharmaceuticals (e.g., strontium, samarium) within 8 weeks of receiving cyclophosphamide on Day -3
5. Has untreated or uncontrolled CNS metastases, including patients who require glucocorticoid therapy for CNS metastases
6. Has received prior treatment with ONT-10 or varlilumab, or prior treatment with other MUC1 vaccines or CD27-targeted agents
7. Has active autoimmune disease or a documented history of autoimmune disease, or history of potential autoimmune syndrome that required systemic steroids or immunosuppressive medications, except for patients with vitiligo, endocrinopathies, type 1 diabetes, or patients with resolved childhood asthma/atopy or other syndromes which would not be expected to recur in the absence of an external trigger (e.g., drug-related serum sickness or post-streptococcal glomerulonephritis). Patients with mild asthma who require intermittent use of bronchodilators (such as albuterol) who have not been hospitalized for asthma in the preceding 3 years will not be excluded from this study.
8. Has recognized immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia, and/or other hereditary congenital immunodeficiencies
9. Has any pre-existing medical condition requiring systemic chronic steroid or immunosuppressive therapy

   a) Inhaled corticosteroids for COPD or topical steroids are allowed
10. Known to be positive for HIV, or to have active hepatitis B, or hepatitis C, or have active infection of any kind requiring systemic therapy
11. Administration of any other vaccine ≤ 4 weeks of receiving cyclophosphamide on Day -3
12. Underlying medical condition that, in the Investigator's opinion, will make the administration of study treatment hazardous or obscure the interpretation of toxicity determination of adverse events. This includes other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancer; or any other cancer from which the patient has been disease-free for at least 3 years.
13. Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension (persistent systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications) or arrhythmia, congestive heart failure (NYHA Class III or IV) related to primary cardiac disease, ischemic or severe valvular heart disease, or myocardial infarction within 6 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Cycles of 12 weeks
  Assessment of the adverse event profile as an indication of overall safety and tolerability of the combination treatment with ONT-10 and varlilumab

SECONDARY OUTCOMES:
Immune Response to MUC1 | 8 weeks on a weekly basis, followed by every 6 weeks
  Determine the immune response of the drug combination of varlilumab and ONT-10 to MUC1 specific humoral and cellular responses.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of Colorado, Aurora, Colorado
  - NYU Perlmutter Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee